CLINICAL TRIAL: NCT01404130
Title: A Pilot Study of the Effects of Isotretinoin on Cognition, Learning and Memory
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Dr Anthony D Ormerod Principal Investigator, University of Aberden
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07/S0802/135
Record Dates: First submitted 2011-07-19; First posted 2011-07-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Acne Vulgaris
Keywords: isotretinoin; hippocampus; memory; learning; CANTAB
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isotretinoin therapy (Experimental): 0.5-1mg /kg titrated by clinical need and tolerance of each patient according to normal clinical practice
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — 0.5-1mg/kg daily for 4-6 months
  Other Names: Accutane, Roaccutane, 13-cid retinoic acid

SUMMARY:
This prospective study tested the effects of isotretinoin in a cohort of patients receiving standard therapy for acne vulgaris. Subjects completed questionnaires and standardised computer based cognitive testing using CANTAB to test for cognitive effects particularly on learning and memory. Test were conducted before starting isotretinoin, after 3 months and again a month after finishing therapy. This was carried out as a pilot study to

1. Test the hypothesis that oral isotretinoin, over its 4-month treatment time, will result in a decline in learning and memory as measured using the CANTAB series of test.
2. Generate data for sample size calculation for a larger study to determine the changes in memory over time in drug and control group
3. Test of CANTAB, questionnaires and data collection forms
4. Select most appropriate outcome measures
5. Identify therapy sensitive cognitive tasks which would be used in future functional brain imaging studies It was not considered to randomise subjects to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects age 16 and over with acne vulgaris
2. Cases should be candidates for isotretinoin therapy should have severe acne not responding to treatment and at risk of scarring and have discussed the risks, pregnancy prevention program and benefits of this treatment according to normal clinical practise

Exclusion Criteria:

1. Subjects already on treatment with isotretinoin
2. Subjects with below normal intelligence who would not understand the CANTAB psychological tests
3. Subjects with neurological disease e.g. epilepsy or pre-existing mental health problems
4. Pregnant females or females not taking preventive precautions
5. Subjects on sedative or psycho-active medications that could interfere with the outcomes tested

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Cognitive change measured by delayed matching to sample (CANTAB) | 3 months on treatment

SECONDARY OUTCOMES:
Change in spacial recognition memory (CANTAB) | 0, 3 months and one month after stopping
Change in Paired Associate learning (CANTAB) | 0, 3 months and one month after stopping
Change in Spacial recognition memory | 0, 3months and one month after stopping
Cambridge gambling task - changes | 0, 3months and one month after stopping

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Ormerod, MB MD FRCP, Principal Investigator — University of Aberdeen
Locations (1):
- Anthony Ormerod, Aberdeen, Aberdeenshire, United Kingdom